CLINICAL TRIAL: NCT03064282
Title: Treatment of Prostatic Hyperplasia With Topical Papaverine
Brief Title: Prostatic Hyperplasia Treatment and Cancer Prevention
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Manchanda Medical Clinic (Other)
Responsible Party: Principal Investigator, DR. VINOD C TAWAR, Principal Investigator, Manchanda Medical Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Tawar - 2
Record Dates: First submitted 2016-12-12; First posted 2017-02-27 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Papaverine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Drug free base as placebo
  Interventions: Other: Placebo
- group two- papaverine arm (Experimental): papaverine in a suitable base
  Interventions: Drug: papaverine

INTERVENTIONS:
Other: Placebo — observation of skin changes if any
  Other Names: drug free base
  Arms: Placebo
Drug: papaverine — observation of symptoms
  Arms: group two- papaverine arm

SUMMARY:
Treatment of patients with prostatic hyperplasia with topical papaverine.

DETAILED DESCRIPTION:
Patients with obstructive voiding and high PSA to be studied for the regression of symptoms and declining PSA.

ELIGIBILITY:
Inclusion Criteria:

* patients with symptoms e.g. obstructive voiding, hyperplasia and high PSA

Exclusion Criteria:

* patients on chemotherapy
* abnormal lab values e.g. liver function, GFR and CAD

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-06-30 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Laboratory tests to measure regression of symptoms | every 4 weeks up to 16 weeks
  patients follow-up on regular intervals

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hafez B, Hafez ES. Andropause: endocrinology, erectile dysfunction, and prostate pathophysiology. Arch Androl. 2004 Mar-Apr;50(2):45-68. PMID 14761837